CLINICAL TRIAL: NCT05219916
Title: Selection of Farnesoid X Receptor (FXR) Ligands as Latency Reversal Agents (LRA) of Latent HIV Proviruses in Circulating CD4+ T Lymphocytes Isolated From Patients With Undetectable HIV Viremia Under cART (Combined Antiretroviral Treatments)
Brief Title: Selection of Farnesoid X Receptor (FXR) Ligands on the Reactivation of Latent HIV Proviruses
Acronym: FXR#2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It is unlikely that the scientific question will ever be answered. Thus, it would be considered unethical to continue the trial.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL21_0846
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Human Immunodeficiency Virus I Infection
Keywords: HIV; LRA; FXR; Reactivation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Descriptive physiopathological study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients infected by HIV, controlled under treatment. (Experimental): Blood sample collection from HIV controlled patients during their scheduled consultation, after obtaining their non-opposition by an investigator.
  Interventions: Procedure: Blood collection.

INTERVENTIONS:
Procedure: Blood collection. — One additional 80 mL blood collection will be collected from HIV patients during a scheduled blood collection as part of their regular follow-up.
  Samples will be transported within 3-5 hours by a carrier approved for the transportation of infectious biological samples from the Croix Rousse hospital to the P3 laboratory of the Ecole Normale Supérieure, Lyon for analysis.

SUMMARY:
The FXReservoir#1 study (NCT03618862) showed that certain FXR ligands reactivate latent viruses in the reservoir circulating in all HIV+ patients tested. These molecules appear as latency reversal agents (LRA) of silent viruses of the HIV reservoir. They can be part of the strategy to eradicate this reservoir, responsible for recurrences of the infection when combined anti-retroviral treatments are stopped.

Two effective leads have been identified on in vitro tests and on ex vivo reactivation using FXReservoir#1. These molecules come from a chemical library of FXR ligands developed by the Inserm team behind the discovery of a role for FXR in viral infections.

A first series of optimized molecules derived from these leads has been synthesized; these molecules, after screening on viral and ADMET (Absorption, Distribution, Metabolisme, Excretion and Toxicity) in vitro tests, must be tested ex vivo on CD4+ lymphocytes from the circulating peripheral reservoir of HIV+ patients in order to select the best molecules with LRA activity. This step is essential before considering the clinical development of an LRA.

ELIGIBILITY:
Inclusion Criteria:

* Criteria relating to the population studied: patients aged 18 to 65 years old, men or women, regardless of ethnic origin.
* Nosological criteria: HIV-1 infection, documented by a complete western blot and/or a detectable viral load at the time of diagnosis, regardless of the viral subtype.
* Pathology severity and progression criteria: patients with a CD4+ count greater than 500 elements/mm3 at the last follow-up visit prior to inclusion in the study. Undetectable viral load for at least six months on stable treatment.
* Criteria relating to treatments/strategies/procedures: Current cART treatment mandatory, regardless of the combination of anti-retrovirals, effective with undetectable viral load. The number of processing lines is not limited.
* Criteria relating to regulation: Absence of opposition

Exclusion Criteria:

* Criteria relating to the population studied: pregnant or breastfeeding women
* Criteria relating to contraindications to the protocol explorations:

Acute or chronic anaemias Acute infections, fever Coagulation disorders, patients taking anticoagulants

- Criteria relating to regulation: Subjects placed under judicial safeguard, guardianship or curatorship Subjects participating in another research with an ongoing exclusion period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Measurement of the reactivation level and the EC50 of the optimized molecules. | At inclusion.
  Measurement of reactivation level compared to that obtained with the reference LRA Ingenol, and EC50 of molecules derived from active leads and preselected on viral and ADMET criteria in vitro to allow the choice of the best molecule for future clinical development.
  PBMCs (peripheral blood mononuclear cells) and rCD4+Tcells will be isolated and treated with the test molecules for 3 days. The treated cells will be incubated to determine the number of cells producing HIV/ million of rCD4+ T cells. FXR ligands will be used at 10 µM. Dose-response assay will be carried out to determine the EC50 (half maximal effective concentration) of the active molecules and the best molecules in the final selection will be tested in combination with inhibitors of the metabolic pathway to confirm their specificity of action.
  Molecules derived from the 2 leads will be screened in successive series.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan FERRY, MD-PhD, Principal Investigator — Service des maladies infectieuses et tropicales, Hôpital de la Croix Rousse, Hospices Civils de Lyon
Locations (1):
- Service des maladies infectieuses et tropicales Hôpital de la Croix Rousse, Lyon, France